CLINICAL TRIAL: NCT04869826
Title: Calibration of the Cloud DX Pulsewave Health Monitor (PAD-2A) Oscillometric Wrist Cuff Home Blood Pressure Monitor, According to the AAMI/ESH/ISO Universal Standard (ISO 81060-2: AMD_2020) (CCV-4)
Brief Title: Calibration of a Wrist Cuff Blood Pressure Device, According to the AAMI/ESH/ISO Universal Standard
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cardiovascular Research New Brunswick (Other)
Collaborators: Cloud DX Inc. (Industry); Horizon Health Network (Other); New Brunswick Health Research Foundation (Other); Dalhousie University (Other)
Responsible Party: Sponsor
Other Study IDs: RS#: 2021-3003; R#: 101246; STP-PW2-002 (Other: Health Canada)
Record Dates: First submitted 2021-04-28; First posted 2021-05-03 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure; Telemedicine; Telemonitoring; Vital sign monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Outpatients Complicated Hypertension Clinic: This study population consists of approximately 200 adult male and female participants (≥ 19 years of age; minimum 30% male/female). Participants will be recruited from eligible patients who are referred to the Complicated Hypertension Clinic at the Saint John Regional Hospital (SJRH) as well as non-patient participants who are willing to volunteer to consent to participate in the study.
  Interventions: Device: Pulsewave Health Monitor (PAD-2A) Device

INTERVENTIONS:
Device: Pulsewave Health Monitor (PAD-2A) Device — This is an observational, comparison study of blood pressure measurements. The objective of this study is to calibrate the blood pressure measurements of the Pulsewave Health Monitor (PAD-2A) device to be within 5±8 mmHg of the average of the dual-observer auscultatory blood pressure measurements via an aneroid sphygmomanometer (reference device), as per the ISO 81060-2: AMD_2020 universal protocol.

SUMMARY:
The objective of this study is to calibrate the blood pressure measurements of the Pulsewave Health Monitor (PAD-2A) device to be within 5±8 mmHg of the average of the dual-observer measurements via an aneroid sphygmomanometer (reference device), as per the methodology described in the ISO 81060-2: AMD_2020 protocol.

DETAILED DESCRIPTION:
The plan for this study is to calibrate the blood pressure measurements of the PAD-2A device with the dual-observer blood pressure measurements via an aneroid sphygmomanometer (reference device), as per the ISO 81060-2: AMD_2020 protocol. The data will be collected and analyzed in order to calibrate the PAD-2A device blood pressure measurements to be within 5±8 mmHg of the average of the dual-observer auscultatory blood pressure measurements by adjusting the device algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 19 years of age (minimum 30% male/female)
* Wrist circumference between 13.5 cm. - 23 cm. (5.3 in. - 9.1 in.):

Specifically for this test device, the wrist size of the consented participants will be distributed accordingly for a Gaussian distribution:

Lowest Octile: ≥ 13.5cm to < 14.7cm Lower Quarter: ≥ 13.5cm to < 15.9cm Lower-Middle Quarter: ≥ 15.9cm to < 18.3cm Upper-Middle Quarter: ≥ 18.3cm to < 20.7cm Upper Quarter: ≥ 20.7cm to ≤ 23.0cm Highest Octile: ≥ 21.9cm to ≤ 23.0cm

● Willing to volunteer to participate and to sign the study specific informed consent form

Exclusion Criteria:

* Wrist circumference less than 13.5 cm. (5.3 in.) or greater than 23 cm. (9.1 in)
* Hand or body tremors
* Irregular heart rhythm (bigeminy, trigeminy, isolated ventricular premature beat (VPB), atrial fibrillation)
* Korotkoff sound K5 not audible
* Pregnant
* A musculoskeletal disorder that prevents a non-invasive device to be inflated/deflated on the arm
* Unwilling to volunteer to participate and to sign the study specific informed consent form

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For this study, we will recruit and consent approximately 200 adult male and female patient participants (≥ 19 years of age; minimum 30% male/female) who are referred to the Complicated Hypertension Clinic at the Saint John Regional Hospital (SJRH) and non-patient participants who are willing to volunteer to consent to participate in the study. Eligibility of participants for this study is based on the inclusion and exclusion criteria as per the ISO 81060-2: AMD_2020 protocol, as described below.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Systolic Pressure | From the start of cuff inflation to the end of cuff deflation (approximately 60 seconds)
  Non-invasive Pulsewave Health Monitor (PAD-2A) wrist cuff blood pressure device (mmHg)
Systolic Pressure | From the start of manual inflation of the upper arm blood pressure cuff to the end of (manual) deflation of the upper arm blood pressure cuff (approximately 30-60 seconds)
  Simultaneous auscultatory blood pressure measurements by 2 trained observers
Diastolic Pressure | From the start of cuff inflation to the end of cuff deflation (approximately 60 seconds)
  Non-invasive Pulsewave Health Monitor (PAD-2A) wrist cuff blood pressure device (mmHg)
Diastolic Pressure | From the start of manual inflation of the upper arm blood pressure cuff to the end of (manual) deflation of the upper arm blood pressure cuff (approximately 30-60 seconds)
  Simultaneous auscultatory blood pressure measurements by 2 trained observers

CONTACTS AND LOCATIONS:
Overall Officials: Martin MacKinnon, MD, FRCP(C), Principal Investigator — Complicated Hypertension Clinic, Saint John Regional Hospital
Locations (1):
- Horizon Health Network, Saint John, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Currently, the clinical research group is undecided regarding individual participant data (IDP) sharing with other researchers upon completion of this study, although it is acknowledged that the practice of data sharing among scientists, clinicians, and other professionals is of increasing importance, particularly for transparency in clinical research studies.

REFERENCES:
- See also: Cloud DX device company website. — https://clouddx.com/